CLINICAL TRIAL: NCT06768515
Title: ICU Management of Brain-Dead Donors Before Multi-Organ Procurement and Factors Associated With the Number of Organs Retrieved
Acronym: DONOR-OBS
Status: Recruiting | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-04
Record Dates: First submitted 2024-12-23; First posted 2025-01-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Death, Brain
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Organ donation: Patients over 18 years of age, hospitalized in the ICU In a state of brain death No objection to organ donation during their lifetime
  Interventions: Other: No interventtion

INTERVENTIONS:
Other: No interventtion — to enhance the understanding of the factors associated with the number of organs retrieved from patients admitted to the ICU for organ donation

SUMMARY:
Solid organ transplantation is the treatment of choice for end stage organ failure to improve patients' quality of life and survival. Each year, more than 5,000 solid organ transplants are performed in France, mainly from brain death donors (BDD).

Approximately 1,500 BDD donors have one or more organs removed each year. Despite the growing demand for transplanted organs, the number of organs available from deceased donors has remained stable over the past few decades. This highlights the need to optimize the management of potential BDD, in order to increase both the quality and number of transplanted organs. Several studies have found an association between the characteristics and management of BDD donors and the number of organs, or even the function of transplanted organs. Data suggest that hemodynamic, respiratory, and metabolic therapeutic targets during BDD management prior to multi-organ procurement were associated with a higher number of transplanted organs compared to standard care. However, this has never been confirmed in a French population. Furthermore, while the impact of these therapeutic goals has been studied after the donor is in a state of brain death, the events occurring in the ICU before reaching brain death status and their impact on the number of organs retrieved have not been investigated. Lastly, the intensity of the therapeutic interventions used to achieve these goals, and certain management delays, have only been partially studied.

Our hypothesis is that achieving a bundle of therapeutic goals, and the intensity of the interventions used to reach these goals, both before and after BDD, are associated with a greater number of organs retrieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, hospitalized in the ICU
* In a state of brain death
* No objection to organ donation during their lifetime
* Patients with social security coverage

Exclusion Criteria:

* Objection to the use of their data during their lifetime
* Registration in the national refusal registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in a state of brain dead. Patients meeting the inclusion criteria from January 1, 2022, to December 31, 2024, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure | Between admission to intensive care and brain death and before multi-organ retrieval
  Mean arterial pressure (MAP) between 60 and 110 mmHg
Central venous pressure | Within 7 last days before brain death and before multi-organ retrieval
  Central venous pressure (CVP) between 4 and 12 mmHg
Left ventricular ejection fraction | Between admission to intensive care and brain death and before multi-organ retrieval
  Left ventricular ejection fraction (LVEF) ≥ 50%
vasopressor | Between admission to intensive care and brain death and before multi-organ retrieval
  Low doses and a single vasopressor. (≤10 µg/kg/min of dopamine or ≤60 µg/min of Neosynephrine or ≤10 µg/min of norepinephrine))
Arterial pH | Between admission to intensive care and brain death and before multi-organ retrieval
  Arterial pH between 7.3 and 7.5
PaO2/FiO2 | Between admission to intensive care and brain death and before multi-organ retrieval
  PaO2/FiO2 ≥ 300
Sodium levels | Between admission to intensive care and brain death and before multi-organ retrieval
  Sodium levels ≤ 155 mmol/L
Diuresis | Between admission to intensive care and brain death and before multi-organ retrieval
  Diuresis ≥ 0.5 mL/kg/h
Blood glucose | Between admission to intensive care and brain death and before multi-organ retrieval
  Blood glucose ≤ 1.5 g/L

SECONDARY OUTCOMES:
demographics of Brain dead | Between admission to intensive care and brain death and before multi-organ retrieval
  The demographics of Brain dead
Causes of neurological injury leading to brain death | Between admission to intensive care and brain death and before multi-organ retrieval
  Describe the causes of neurological injury leading to brain death
Timelines and durations of patient management before and after brain death | Between admission to intensive care and brain death and before multi-organ retrieval
  Descibe the timelines and durations of patient management before and after brain death
Incidence of organ failures before and after brain death | Between admission to intensive care and brain death and before multi-organ retrieval
  Describe the incidence of organ failures before and after brain death
Incidence of acute kidney failure before and after brain death | Between admission to intensive care and brain death and before multi-organ retrieval
  Describe the incidence of acute kidney failure before and after brain death
Incidence of infections, sepsis, and septic shock before and after brain death | Between admission to intensive care and brain death and before multi-organ retrieval
  Describe the incidence of infections, sepsis, and septic shock before and after brain death
Incidence of diabetes insipidus | Between admission to intensive care and brain death and before multi-organ retrieval
  Describe the incidence of diabetes insipidus
Treatments administered before and after brain death | Between admission to intensive care and brain death and before multi-organ retrieval
  Describe the treatments administered before and after brain death
Number and nature of organs retrieved | Between admission to intensive care and brain death and before multi-organ retrieval
  Describe the number and nature of organs retrieved, including heart, lungs (2 organs), kidneys (2 organs), liver, pancreas
Number and nature of organs available for transplantation | Between admission to intensive care and brain death and before multi-organ retrieval
  Describe the number and nature of organs available for transplantation, including heart, lungs (2 organs), kidneys (2 organs), liver, pancreas
Number of organs placed on ex situ preservation and the type of preservation method used | Between admission to intensive care and brain death and before multi-organ retrieval
  Describe the number of organs placed on ex situ preservation and the type of preservation method used
Number, causes, and associated factors of unsuccessful organ retrieval procedures | Between admission to intensive care and brain death and before multi-organ retrieval
  Desctibe the number, causes, and associated factors of unsuccessful organ retrieval procedures

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Saint-Louis, AP-HP, Paris
  - Hôpital Pitié Salpêtrière AP-HP, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malinoski DJ, Patel MS, Daly MC, Oley-Graybill C, Salim A; UNOS Region 5 DMG workgroup. The impact of meeting donor management goals on the number of organs transplanted per donor: results from the United Network for Organ Sharing Region 5 prospective donor management goals study. Crit Care Med. 2012 Oct;40(10):2773-80. doi: 10.1097/CCM.0b013e31825b252a. PMID 22846779
- [Background] Oniscu GC, Rockell K, Martin DE. Challenges in undertaking research in transplantation. Lancet. 2025 Mar 1;405(10480):681-683. doi: 10.1016/S0140-6736(24)00931-0. Epub 2024 May 21. No abstract available. PMID 38788740
- [Background] iomedecine, P. Chiffres 2022 de l'activité de prélèvement et de greffe d'organes et de tissus et Baromète 2023 sur la connaissance et la perception du don d'organes en France.
- [Result] Patel MS, De La Cruz S, Sally MB, Groat T, Malinoski DJ. Active Donor Management During the Hospital Phase of Care Is Associated with More Organs Transplanted per Donor. J Am Coll Surg. 2017 Oct;225(4):525-531. doi: 10.1016/j.jamcollsurg.2017.06.014. Epub 2017 Jul 21. PMID 28739153
- [Result] Bera KD, Shah A, English MR, Harvey D, Ploeg RJ. Optimisation of the organ donor and effects on transplanted organs: a narrative review on current practice and future directions. Anaesthesia. 2020 Sep;75(9):1191-1204. doi: 10.1111/anae.15037. Epub 2020 May 19. PMID 32430910
- [Result] Patel MS, Zatarain J, De La Cruz S, Sally MB, Ewing T, Crutchfield M, Enestvedt CK, Malinoski DJ. The impact of meeting donor management goals on the number of organs transplanted per expanded criteria donor: a prospective study from the UNOS Region 5 Donor Management Goals Workgroup. JAMA Surg. 2014 Sep;149(9):969-75. doi: 10.1001/jamasurg.2014.967. PMID 25054379